CLINICAL TRIAL: NCT00095134
Title: A Double-Blind Study Comparing Adjunctive Risperidone Versus Placebo in Major Depressive Disorder That Is Not Responding to Standard Therapy
Brief Title: Study Comparing Adjunctive Risperidone Versus Placebo in Major Depressive Disorder That Is Not Responding to Standard Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Janssen, LP (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR004726
Record Dates: First submitted 2004-11-01; First posted 2004-11-01 (Estimated); Last update posted 2011-12-06 (Estimated); Status verified 2011-12

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Risperidone

INTERVENTIONS:
Drug: risperidone

SUMMARY:
The purpose of this trial is to evaluate the efficacy and safety of risperidone versus placebo in subjects with Major Depressive Disorder with sub-optimal response to antidepressant therapy.

DETAILED DESCRIPTION:
Many patients who suffer from Major Depressive Disorder (MDD) do not benefit or show only partial benefit from current psychotropic therapy. This clinical trial seeks to study the efficacy and safety of adjunctive treatment with risperidone in patients with MDD who failed to adequately respond to standard antidepressant treatment prior to this trial and who prospectively do not respond to adequate treatment with standard antidepressant therapy (SAD).

Patients entering the open label phase of the study will have already taken a commercially available SAD for a minimum of 4 weeks, and provided the dose was optimal, will continue on this dose of SAD throughout the four-week open-label and six-week double-blind phases of the trial.

If the dose in the four weeks prior to entering the study was not optimal (as per standard clinical practice), the dose will be increased to be within the optimal range and continued at that dose through the entire open-label SAD and double-blind phases.

During the double-blind phase, subjects receive an adjunctive dose of risperidone or placebo, once daily, added to their stable dose of SAD. The starting dose of risperidone or placebo is 0.25 mg for the first three days of the double-blind phase, and is increased to 0.5 mg for days 4 through 14. On the 15th day of this phase, the dose is increased to the target dose of 1.0 mg/day. If response to this dose is not optimal by day 29, it is increased to 2.0 mg/day and is maintained for the duration of the 6-week double-blind phase. This dose may be reduced once to 1.0 mg/day, but then must be maintained at that dose for the remainder of the study.

ELIGIBILITY:
Inclusion Criteria:

* Understand and sign the informed consent form
* Age 18-65
* Healthy on the basis of Physical Exam
* Treatment with a single antidepressant 4 weeks prior to study start and willingness to maintain on stable dose of the same antidepressant throughout the study
* Current diagnosis of Major Depressive Disorder
* Judgement of the clinician that the subject has shown a sub-optimal response to the antidepressant

Exclusion Criteria:

* Presence of other serious medical illness(es)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 630 (Actual)
Dates: Start 2004-10; Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Difference in therapeutic effect of risperidone and placebo as measured by change in depression rating scale (HAM-D) at end of week 4 of the double-blind phase.

SECONDARY OUTCOMES:
Safety will be assessed through reported adverse events and vital signs (weight, blood pressure, pulse, and temperature).

CONTACTS AND LOCATIONS:
Locations (70):
- United States (70):
  - Innovative Clinical Trials, LLC, Birmingham, Alabama
  - Greystone Medical Research, Birmingham, Alabama
  - Scottsdale Family Health, Scottsdale, Arizona
  - Sun Valley Medical, Sun City, Arizona
  - Southwest Biomedical Research Foundation, Tucson, Arizona
  - Southwestern Research Institute, Burbank, California
  - Chrishard Clinical Research, Inglewood, California
  - Optimum Health Services, La Mesa, California
  - Pacific Insititute for Medical Research, Los Angeles, California
  - Optimum Health Services, Oceanside, California
  - Behavioral Health 2000, LLC, Riverside, California
  - nTouch Research, San Diego, California
  - Psychiatric Medicine Center, New London, Connecticut
  - Glasgow Family Practice, Newark, Delaware
  - Leonard Bass, MD, PA, Fort Lauderdale, Florida
  - Sarkis Clinical Trials, Gainesville, Florida
  - Roger Miller, MD, Jacksonville, Florida
  - BioQuan Research Group, Inc., North Miami, Florida
  - Family Practice - St. Cloud, Saint Cloud, Florida
  - Allan B. Aven, MD, Arlington Heights, Illinois
  - nTouch Research - Chicago, Naperville, Illinois
  - nTouch Research - Peoria, Peoria, Illinois
  - Balanced Health Research Center, Peoria, Illinois
  - American Health Network, Avon, Indiana
  - Research Solutions - Evansville, Evansville, Indiana
  - Amy Kaissar, MD, Indianapolis, Indiana
  - Clinco, Terre Haute, Indiana
  - Hartford Research Group, Florence, Kentucky
  - New Orleans Medical Institute, Metairie, Louisiana
  - Brentwood Research Institute, Shreveport, Louisiana
  - Professional Clinical Research at Great Lakes Family Care, Cadillac, Michigan
  - Sam Hawatmeh, MD, PC, St Louis, Missouri
  - Alliance Medical Center, PC, Alliance, Nebraska
  - Clinical Trial Associates, Glendora, New Jersey
  - Partners in Primary Care, Turnersville, New Jersey
  - ABQ Med., P.C., Albuquerque, New Mexico
  - Eastside Comprehensive Medical Services, LLC, New York, New York
  - Raleigh Medical Group, Raleigh, North Carolina
  - Salem Research Group, Winston-Salem, North Carolina
  - Community Health Care, Inc., Canal Fulton, Ohio
  - Community Research Management Associates, Inc., Cincinnati, Ohio
  - Hightop Medical Research Center, Cincinnati, Ohio
  - CFP Research, Inc., Cincinnati, Ohio
  - Martin Schear, MD, Dayton, Ohio
  - Family Practice Center of Wadsworth, Wadsworth, Ohio
  - Sooner Clinical Research, Edmond, Oklahoma
  - Med-line Research, Moore, Oklahoma
  - Cutting Edge Research Group, Oklahoma City, Oklahoma
  - Advanced Clinical Trials, Eugene, Oregon
  - Clinical Research Consultants/Providence Medical, Medford, Oregon
  - Medford Medical Clinic, LLP, Medford, Oregon
  - Gateway Medical, Downingtown, Pennsylvania
  - Feasterville Family Health Care, Feasterville, Pennsylvania
  - Detweiler Family Medicine, Lansdale, Pennsylvania
  - Green & Seidner Family Practice, Lansdale, Pennsylvania
  - Woodburne Family Practice, Levittown, Pennsylvania
  - Pearl Clinical Research, Norristown, Pennsylvania
  - Joseph Rybicki, MD, Philadelphia, Pennsylvania
  - Clinical Trials Research Services, LLC, Pittsburgh, Pennsylvania
  - Consolidated Clinical Trials, Inc., Pittsburgh, Pennsylvania
  - Charles Buttz, MD, Pottstown, Pennsylvania
  - Research Across America, Reading, Pennsylvania
  - The Family Practice, Greer, South Carolina
  - Harmony Clinical Research, Johnson City, Tennessee
  - DiscoveResearch, Inc., Beaumont, Texas
  - South Texas Applied Research, Corpus Christi, Texas
  - International Clinical Research Associates, LLC, Richmond, Virginia
  - International Clinical Research Associates, Virgina Beach, Virginia
  - Richard Neiman, MD, Kirkland, Washington
  - Daniel Blizzard, MD, Spokane, Washington

REFERENCES:
- [Derived] Pandina G, Turkoz I, Bossie C. Impact of self-reported juvenile abuse on treatment outcome in patients with major depressive disorder. J Affect Disord. 2013 Oct;151(1):384-91. doi: 10.1016/j.jad.2013.01.053. Epub 2013 Jul 10. PMID 23849714
- [Derived] Mahmoud RA, Pandina GJ, Turkoz I, Kosik-Gonzalez C, Canuso CM, Kujawa MJ, Gharabawi-Garibaldi GM. Risperidone for treatment-refractory major depressive disorder: a randomized trial. Ann Intern Med. 2007 Nov 6;147(9):593-602. doi: 10.7326/0003-4819-147-9-200711060-00003. PMID 17975181